CLINICAL TRIAL: NCT02588820
Title: Impact of Extremely Early Antiretroviral Therapy to Reduce VIral REservoir and Induce Functional CURE of HIV-1 Infection: A Pilot Comparative Study
Brief Title: Impact of Extremely Early Antiretroviral Therapy to Reduce VIral REservoir and Induce Functional CURE of HIV-1 Infection
Acronym: VIRECURE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: David Garcia Cinca (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor-Investigator, David Garcia Cinca, Clinical Research Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-000251-24
Record Dates: First submitted 2015-10-20; First posted 2015-10-28 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antiretroviral treatment (Experimental)
  Interventions: Drug: Antiretroviral Therapy (Experimental)

INTERVENTIONS:
Drug: Antiretroviral Therapy (Experimental) — 1. Initial ART until HLA-B5701 results became available (48 hours):
     1. Tenofovir 245 mg once a day
     2. Emtricitabine 200 mg once a day
     3. Dolutegravir 50 mg once a day
     4. Darunavir 800 mg once a day
     5. Ritonavir 100 mg once a day
     6. Maraviroc 150 mg twice a day
  2. Three months continuation treatment (after HLA-B5701 confirmed as negative):
     1. Dolutegravir 50 mg once a day.
     2. Abacavir 600 mg once a day
     3. Lamivudine 300 mg once a day
     4. Darunavir 800 mg once a day
     5. Ritonavir 100 mg once a day
     6. Maraviroc 150 mg twice a day The whole treatment schedule comprises 7 pills per day (in a single dose), except for maraviroc, which will be given twice daily.
  3. Nine months continuation treatment (till complete 12 months treatment):
     1. Abacavir, 600mg once a day
     2. Lamivudine, 300 mg once a day
     3. Dolutegravir, 50 mg once a day

SUMMARY:
Pilot study to evaluate the impact of extremely early ART in the dynamics of viral reservoir, immune activation and inflammation in patients with HIV-1 infection of less than 20 days (Fiebig stages I-II) compared to patients with infection of 20-100 days (Fiebig stages III-V), to induce HIV functional cure.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men
* Male's between18 and 65 years old
* Less than 100 days of infection
* Patient stage Fiebig I to V
* Negative or Incomplete western blot with negative p31 band

Exclusion Criteria:

* P31 positive band in western blot
* Positive Delta32 CCR5 mutation, HLA-B5701 or HLA-B27 (´late' exclusion criteria)
* Active oncological disease
* Active hepatitis C virus infection

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Functional cure (Proportion of patients with undetectable viral reservoir) | 12 months of treatment
  Proportion of patients in both groups with undetectable viral reservoir in peripheral and rectal tissue CD4+ T cells. A viral load will be performed at 1, 3 and 12 months after ART initiation and in rectal tissue at one year post-ART initiation.

SECONDARY OUTCOMES:
Proportion of patients with undetectable plasmatic HIV viral load | 1, 3 and 12 months post-stop antiretroviral treatment will be evaluated.
  In those patients with undetectable viral reservoir stopping antiretroviral treatment at 12 months
Level of reduction of viral reservoir among patients treated in phase I-II Fiebig and patients treated in Fiebig stage III-V | 1, 3, 12 months will be measured in patients on antiretroviral treatment and at 1, 3, 12 months post-stop
Level of reduction of bacterial translocation among patients treated in phase I-II Fiebig and patients treated in Fiebig stage III-V | 1, 3, 12 months will be measured in patients on antiretroviral treatment and at 1, 3, 12 months post-stop
Level of reduction of immune activation among patients treated in phase I-II Fiebig and patients treated in Fiebig stage III-V | 1, 3, 12 months will be measured in patients on antiretroviral treatment and at 1, 3, 12 months post-stop
Level of reduction of inflammation among patients treated in phase I-II Fiebig and patients treated in Fiebig stage III-V | 1, 3, 12 months will be measured in patients on antiretroviral treatment and at 1, 3, 12 months post-stop

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic i Provincial de Barcelona, Barcelona, Barcelona, Spain